CLINICAL TRIAL: NCT06510205
Title: Post-Market Clinical Follow-up for Mentor Breast Implants
Brief Title: The Study is an Oberservational Post-market Follow-up Program to Evaluate Long Term(5 Years) Safety of Mentor Breast Implants in Chinese Population.
Status: Recruiting | Type: Observational
Sponsor: Johnson & Johnson Medical (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MNT202401; MNT202401 (Other: Johnson & Johnson Medical (Shanghai) Ltd)
Record Dates: First submitted 2024-07-05; First posted 2024-07-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Breast Augmentation and Breast Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mentor Group: Who recieves Mentor breast implants per request
  Interventions: Device: Mentor Breast implants

INTERVENTIONS:
Device: Mentor Breast implants — Mentor breast implants are circular or waterdrop-shaped devices with shells made of successive cross-linked layers of silicone elastomer. The shell is filled with Mentor's proprietary formulation of silicone gel.
  Mentor breast implants are available in smooth and textured shells, both supplied in sterile form.

SUMMARY:
The Mentor Post-Market Clinical Follow-Up Study is a multicenter observational study conducted in China. It aims to collect safety data on Mentor breast implants over a 5-year follow-up period in the Chinese population. In addition to safety data, the study will also gather information on postoperative pain and participant satisfaction levels. The objective is to explore customers' clinical experiences and use them as a reference for future product development. The study intends to enroll a minimum of 300 subjects per license, with participation from three or more medical institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have received Mentor breast implants per product instructions;
2. Participants must possess the ability to comprehend the study procedures, give consent for the use of their preoperative and surgical data, and agree to take part in postoperative follow-up assessments. Additionally, they should possess the necessary civil capacity, be capable of reading and writing, and willingly provide informed consent by signing the consent form.
3. Participants must be at least 22 years old at the time of their implantation surgery.

Exclusion Criteria:

* Not applicable

Ages: 22 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Per product instruction for use(IFU)
Study Population: All populations receiving Mentor breast implants
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2034-06-30 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Breast implant related AEs | Up to 5 years
  Post-op 1 month, 3 months, 1 year, 2 years, 3 years, 4 years, 5 years

SECONDARY OUTCOMES:
Numerical Pain Scale assessment | 1 month after surgery
  Zero means you have no pain, while 10 represents the most intense pain possible.
Customer Satisfaction Score measurement | Up to 5 years after surgery
  Measured at 1 month, 3 months, 1 year, 2 years, 3 years, 4 years, 5 years after surgery Using a 5-point scoring scale, 5 means very satisfied while 1 means very disatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Huimin Wu, Study Director — Shenzhen Junke Medical Cosmetology Clinic
Locations (3):
- China (3):
  - Sichuan Huamei Zixin Medical Aesthetic Hospital, Chengdu
  - Shenzhen Yixing Medical Cosmetology Hospital, Shenzhen
  - Shenzhen Junke Medical Cosmetology Clinic, Shenzhen

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
  .
URL: http://yoda.yale.edu